CLINICAL TRIAL: NCT07299461
Title: Investigation of the Effects of Combined Low-intensity Resistance Exercise With Blood Flow Restriction on Muscle Strength, Pain, and Fear of Movement in Post-operative Meniscus Rehabilitation
Brief Title: Blood Flow Restriction Training After Meniscus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFKAVAK-UUTEZ 01
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Blood Flow Restriction and Low-Intensity Resistance Training; Meniscal Injuries
Keywords: meniscus; knee pain; Blood Flow Restriction; exercise; physiotherapy
MeSH Terms: conditions — Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm ( traditional treatment ) (Active Comparator): The first group underwent traditional physical therapy exercises and physical therapy modalities for the operated lower extremity for 60 minutes a day, three days a week, for eight weeks.
  Interventions: Other: Traditional physical therapy exercises and physical therapy modalities
- Treatment Group ( traditional treatment + BFR-LIRE exercises treatment ) (Experimental): The second group received the same traditional physical therapy modalities and exercises for 60 minutes a day, three days a week, for eight weeks, with an additional 15-minute BFR-LIRE session aimed at increasing the strength of the operated lower extremity and managing pain.
  Interventions: Other: Traditional physical therapy exercises and physical therapy modalities + low-intensity resistance exercise with blood flow restriction (BFR-LIRE)

INTERVENTIONS:
Other: Traditional physical therapy exercises and physical therapy modalities — * NMES for 20 minutes
  * Therapeutic (Continuous) Ultrasound for 6 minutes
  * Cold Pack (CP) for 7 minutes
  * Conventional Physical Therapy Exercises:
  Stretching exercises targeting the quadriceps femoris, hamstrings, and gastrocnemius muscles were performed by the patient for 30 seconds of stretching followed by 30 seconds of rest, for a total of 3 sets. All stretching movements were supervised by a physiotherapist, and each stretch was performed up to the patient's pain threshold.
  Arms: Control Arm ( traditional treatment )
Other: Traditional physical therapy exercises and physical therapy modalities + low-intensity resistance exercise with blood flow restriction (BFR-LIRE) — In addition to the other intervention group procedures, a 15-minute low-intensity resistance exercise program with BFR-which is known to be effective in increasing muscle strength despite being performed at low intensity-was included in the patients' treatment protocol.
  Arms: Treatment Group ( traditional treatment + BFR-LIRE exercises treatment )

SUMMARY:
This study was conducted to investigate the effects of combined low-intensity resistance exercise with blood flow restriction (BFR-LIRE) on muscle strength, pain, and fear of movement in individuals who had undergone post-operative meniscus surgery.

A total of 36 individuals who reported knee pain of 4 or higher on the Visual Analog Scale (VAS) following surgery voluntarily participated in the study. The participants were randomly divided into two groups. The first group underwent traditional physical therapy exercises and physical therapy modalities for the operated lower extremity for 60 minutes a day, three days a week, for eight weeks. The second group received the same traditional physical therapy modalities and exercises for 60 minutes a day, three days a week, for eight weeks, with an additional 15-minute BFR-LIRE session aimed at increasing the strength of the operated lower extremity and managing pain.

Keywords: Pain, Knee Pain, Meniscus, Physiotherapy, Blood Flow Restriction, Exercise

ELIGIBILITY:
Inclusion Criteria:

* Having undergone meniscus repair surgery within the last 6 months
* Being between 20 and 50 years of age
* Being unable to perform high-intensity training
* Having a Visual Analog Scale (VAS) score of 4 or higher

Exclusion Criteria:

* Having a history of hypertension
* Having a history of heart failure or myocardial infarction
* Having a history of Deep Vein Thrombosis (DVT)
* Having Peripheral Artery Disease, varicose veins, or bleeding disorders
* Use of anticoagulants
* Presence or history of peripheral nerve disorders or neuropathy
* History of Diabetes Mellitus
* Having skin sensitivity
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline and after 8 weeks of intervention
  The Visual Analog Scale (VAS) was used to measure the severity of pain felt by the patients in the knee region before and after treatment. VAS is an assessment tool that was first developed in the field of psychology and later began to be used in pharmacology to evaluate pain in rheumatology patients undergoing treatment. Patients are asked to mark the point that indicates their pain intensity on a 100 mm (10-centimeter) scale. An increase in the value indicates that the perceived pain intensity has increased. VAS is a scale that can be administered in a very short time and has high reliability.
Tampa Scale for Kinesiophobia (TSK) | Baseline and after 8 weeks of intervention
  The Tampa Scale for Kinesiophobia (TSK), which is frequently used to assess fear of movement related to pain in individuals with chronic musculoskeletal pain, was preferred in this study to evaluate participants' levels of fear and avoidance associated with movement. The Turkish validity and reliability study of the scale has been conducted. The scale consists of 17 items scored on a Likert scale. Individuals can obtain a score between 17 and 68, and higher scores indicate a greater level of kinesiophobia. Participants were asked to complete the scale themselves by selecting one of the following options for each item: "strongly disagree," "disagree," "agree," or "strongly agree."
Assessment of Range of Motion | Baseline and after 8 weeks of intervention
  While measuring knee flexion and extension angles, patients were positioned supine as recommended by Clarkson et al. In measurements performed using a universal goniometer, the pivot point was placed on the lateral condyle of the femur, the stationary arm was aligned with the lateral midline of the femur, and the movable arm was aligned parallel to the fibula.
Muscle Strength Analysis | Baseline and after 8 weeks of intervention
  Muscle strength measurements were performed using a digital hand-held dynamometer, the "MicroFET2" (Hoggan Health Industries, Draper, UT), which has been shown to be valid and reliable in many studies. Knee extension (quadriceps) muscle strength, knee flexion (hamstring) muscle strength, and ankle plantar flexion (gastrocnemius) muscle strength were measured in accordance with the procedures described in the validity and reliability studies of the MicroFET2 device.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Fatih Kavak, Study Director — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: 09.12.2025-09.12.2026